CLINICAL TRIAL: NCT01090453
Title: Feasibility Study of GlaxoSmithKline Biologicals' GSK2202083A Vaccine in Healthy Infants at 2, 4 and 12 Months of Age
Brief Title: Study of GlaxoSmithKline Biologicals' GSK2202083A Vaccine in Healthy Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 113615
Record Dates: First submitted 2010-03-18; First posted 2010-03-22 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2016-08

CONDITIONS: Tetanus; Hepatitis B; Haemophilus Influenzae Type b; Poliomyelitis; Acellular Pertussis; Diphtheria; Neisseria Meningitidis
MeSH Terms: conditions — Tetanus; Hepatitis B; Haemophilus Infections; Poliomyelitis; Diphtheria | interventions — 13-valent pneumococcal vaccine; diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine; RIX4414 vaccine

ARMS (2):
- GSK2202083A Group (Experimental): Subjects aged between and including 8 and 12 weeks of age at the time of first vaccination received 3 doses of GSK2202083A vaccine, co-administered with Prevenar 13® at 2, 4 and 12 months of age. The GSK2202083A and Prevenar 13® vaccines were administered intramuscularly into the right and left sides of the thigh, respectively. An optional 2-dose vaccination with Rotarix™ was offered to the study participants at 2 and 4 months of age.
  Interventions: Biological: GSK2202083A vaccine; Biological: Prevenar 13®; Biological: Rotarix™
- Infanrix hexa Group (Active Comparator): Subjects aged between and including 8 and 12 weeks of age at the time of first vaccination received 3 doses of Infanrix hexa™ vaccine, co-administered with Prevenar 13® and Menjugate® at 2, 4 and 12 months of age. The Infanrix hexa™ and Prevenar 13® vaccines were administered intramuscularly into the right and upper left sides of the thigh, respectively and the Menjugate® vaccine was administered intramuscularly in the lower left thigh. An optional 2-dose vaccination with Rotarix™ was offered to the study participants at 2 and 4 months of age.
  Interventions: Biological: Prevenar 13®; Biological: Infanrix hexa™; Biological: Menjugate®; Biological: Rotarix™

INTERVENTIONS:
Biological: GSK2202083A vaccine — 3 doses given at 2, 4 and 12 months of age
  Arms: GSK2202083A Group
Biological: Prevenar 13® — 3 co-administered doses
Biological: Infanrix hexa™ — 3 doses given at 2, 4 and 12 months of age
  Arms: Infanrix hexa Group
Biological: Menjugate® — 3 co-administered doses
  Arms: Infanrix hexa Group
Biological: Rotarix™ — Oral, two doses

SUMMARY:
This study will evaluate the safety and immunogenicity of GSK Biologicals' GSK2202083 vaccine co-administered with Prevenar 13® at 2, 4 and 12 months of age and with Rotarix™ at 2 and 4 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parent(s)/Legally Acceptable Representative(s) can and will comply with the requirements of the protocol.
* A male or female infant between, and including, 8 and 12 weeks at the time of the first vaccination.
* Born after a gestation period of 36 to 42 weeks inclusive.
* Written informed consent obtained from the parent(s), Legally Acceptable Representative(s) of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs since birth.
* Child in care.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
* Administration of a vaccine not foreseen by the study protocol within 30 days prior to randomisation, or planned administration from randomisation to the end of the study with the exception of inactivated influenza vaccines. The administration of diphtheria, tetanus, pertussis, hepatitis B, poliomyelitis, Haemophilus influenzae type b, pneumococcal, rotavirus and/or MenC vaccines is not allowed at any time during the study period but other vaccines are allowed during the period from one day after study Visit 3 to 31 days before study Visit 4.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Evidence of previous diphtheria, tetanus, pertussis, hepatitis B, poliomyelitis, Hib, pneumococcal, rotavirus and/or MenC vaccination or disease, including Hepatitis B virus vaccination at birth.
* History of seizures or progressive neurological disease.
* Subjects with history of intussusception or uncorrected congenital malformation of the gastrointestinal tract that would predispose for intussusception.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine(s).
* Major congenital defects or serious chronic illness.

The following condition is temporary or self-limiting, and a subject may be vaccinated once the condition has resolved if no other exclusion criteria is met:

* Current febrile illness or other moderate to severe illness within 24 hours of study vaccine administration.
* Current gastrointestinal infection.

Ages: 8 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 480 (Actual)
Dates: Start 2010-05-17; Primary Completion 2011-10-11 (Actual); Study Completion 2011-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (34):
- Canada (3):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Hamilton, Ontario
- France (9):
  - GSK Investigational Site, Aix-en-Provence
  - GSK Investigational Site, Dax
  - GSK Investigational Site, Draguignan
  - GSK Investigational Site, Essey-lès-Nancy
  - GSK Investigational Site, Floirac
  - GSK Investigational Site, Le Havre
  - GSK Investigational Site, Lingolsheim
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Trélazé
- Germany (22):
  - GSK Investigational Site, Bad Saulgau, Baden-Wurttemberg
  - GSK Investigational Site, Kehl, Baden-Wurttemberg
  - GSK Investigational Site, Schwäbisch Hall, Baden-Wurttemberg
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Tuttlingen, Baden-Wurttemberg
  - GSK Investigational Site, Berchtesgaden, Bavaria
  - GSK Investigational Site, Bindlach, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Nördlingen, Bavaria
  - GSK Investigational Site, Eschwege, Hesse
  - GSK Investigational Site, Wolfenbüttel, Lower Saxony
  - GSK Investigational Site, Detmold, North Rhine-Westphalia
  - GSK Investigational Site, Heiligenhaus, North Rhine-Westphalia
  - GSK Investigational Site, Kleve-Materborn, North Rhine-Westphalia
  - GSK Investigational Site, Löhne, North Rhine-Westphalia
  - GSK Investigational Site, Porta Westfalica, North Rhine-Westphalia
  - GSK Investigational Site, Solingen, North Rhine-Westphalia
  - GSK Investigational Site, Willich, North Rhine-Westphalia
  - GSK Investigational Site, Frankenthal, Rhineland-Palatinate
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Trier, Rhineland-Palatinate
  - GSK Investigational Site, Worms, Rhineland-Palatinate

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 113615 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113615 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113615 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113615 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113615 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113615 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 480 subjects were enrolled in the study.
Period: Overall Study
Arm/Group | GSK2202083A Group | Infanrix Hexa Group
Started | 238 | 242
Completed | 225 | 228
Not Completed | 13 | 14
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 7 | 7
Not completed — Non serious AEs | 1 | 0
Not completed — Protocol Violation | 2 | 0
Not completed — Other | 2 | 4
Not completed — Eligibility Criteria | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK2202083A Group | Infanrix Hexa Group | Total
Number analyzed (Participants) | 238 | 242 | 480
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 9.10 (1.15) | 9.20 (1.17) | 9.15 (1.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 111 | 219
  Male | 130 | 131 | 261
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African heritage/African American | 2 | 3 | 5
  American Indian or Alaskan Native | 2 | 0 | 2
  Asian-Central/South Asian heritage | 1 | 1 | 2
  Asian-East Asian heritage | 5 | 1 | 6
  Asian-South East Asian heritage | 2 | 1 | 3
  White-Arabic/North African heritage | 5 | 8 | 13
  White-Caucasian/European heritage | 210 | 216 | 426
  Unspecified | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Anti-polyribosylribitol Phosphate (Anti-PRP) Above the Cut-off
Description: The anti-PRP antibody concentration cut-off for this assay was greater than or equal to (≥) 0.15 micrograms per milliliter (µg/mL).
Time Frame: At Month 3
Population: The analysis was performed on the According-To-Protocol cohort for immunogenicity, which included all evaluable subjects, who complied with the protocol, for whom immunogenicity data were available and for whom assay results were available for antibodies against at least one study vaccine antigen component at the post-vaccination time points.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A Group | Infanrix Hexa Group
Number analyzed (Participants) | 216 | 223
Participants | 204 | 188

2. Primary Outcome: Number of Subjects With Neisseria Meningitidis Using Baby Rabbit Complement (rSBA-MenC) Antibody Titers Above the Cut-off
Description: The rSBA-MenC antibody titers cut-off for this assay was ≥ 1:8.
Time Frame: At Month 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A Group | Infanrix Hexa Group
Number analyzed (Participants) | 214 | 220
Participants | 210 | 219

3. Secondary Outcome: Number of Subjects With Anti-PRP Antibody Concentrations Above the Cut-offs
Description: The anti-PRP antibody concentration cut-offs for this assay were ≥ 0.15 µg/mL and 1.0 µg/mL. Values concerning the cut-off of 0.15 µg/mL at Month 3 were listed for a primary outcome, hence they were not reported under this outcome.
Time Frame: At Month 3, Month 10 and Month 11.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A Group | Infanrix Hexa Group
Number analyzed (Participants) | 216 | 223
Participants
  Anti-PRP ≥ 1.0, Month 3 | 134 | 82
  Anti-PRP ≥ 0.15, Month 10: number analyzed (Participants) | 197 | 195
  Anti-PRP ≥ 0.15, Month 10 | 145 | 123
  Anti-PRP ≥ 0.15, Month 11: number analyzed (Participants) | 200 | 196
  Anti-PRP ≥ 0.15, Month 11 | 200 | 196
  Anti-PRP ≥ 1.0, Month 10: number analyzed (Participants) | 197 | 195
  Anti-PRP ≥ 1.0, Month 10 | 32 | 26
  Anti-PRP ≥ 1.0 , Month 11: number analyzed (Participants) | 200 | 196
  Anti-PRP ≥ 1.0 , Month 11 | 198 | 185

4. Secondary Outcome: Number of Subjects With rSBA-MenC Antibody Titers Above the Cut-offs
Description: The rSBA-MenC antibody titers cut-off for this assay were ≥ 1:8 and ≥ 1:128. Values concerning the cut-off of 1:8 at Month 3 were listed for a primary outcome, hence they were not reported under this outcome.
Time Frame: At Month 3, Month 10 and Month 11.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A Group | Infanrix Hexa Group
Number analyzed (Participants) | 214 | 220
Participants
  rSBA-MenC ≥ 1:128, Month 3 | 201 | 219
  rSBA-MenC ≥ 1:8, Month 10: number analyzed (Participants) | 194 | 191
  rSBA-MenC ≥ 1:8, Month 10 | 178 | 154
  rSBA-MenC ≥ 1:8, Month 11: number analyzed (Participants) | 199 | 196
  rSBA-MenC ≥ 1:8, Month 11 | 198 | 196
  rSBA-MenC ≥ 1:128, Month 10: number analyzed (Participants) | 194 | 191
  rSBA-MenC ≥ 1:128, Month 10 | 119 | 92
  rSBA-MenC ≥ 1:128, Month 11: number analyzed (Participants) | 199 | 196
  rSBA-MenC ≥ 1:128, Month 11 | 192 | 196

5. Secondary Outcome: Concentrations for Anti-PRP.
Description: Concentrations were expressed as geometric mean concentrations (GMCs). The seroprotection reference cut-off values were ≥ 0.15 µg/mL and ≥ 1.0 µg/mL.
Time Frame: At Month 3, Month 10 and Month 11.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | GSK2202083A Group | Infanrix Hexa Group
Number analyzed (Participants) | 216 | 223
µg/mL
  Anti-PRP at Month 3 | 1.594 [1.306 to 1.946] | 0.671 [0.548 to 0.822]
  Anti-PRP at Month 10: number analyzed (Participants) | 197 | 195
  Anti-PRP at Month 10 | 0.340 [0.283 to 0.407] | 0.260 [0.217 to 0.311]
  Anti-PRP at Month 11: number analyzed (Participants) | 200 | 196
  Anti-PRP at Month 11 | 17.678 [15.058 to 20.753] | 13.737 [11.205 to 16.840]

6. Secondary Outcome: Titers for rSBA-MenC.
Description: Titers were expressed as geometric mean titers (GMCs). The seropositivity reference cut-off values were ≥ 1:8 and ≥ 1:128.
Time Frame: At Month 3, Month 10 and Month 11.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | GSK2202083A Group | Infanrix Hexa Group
Number analyzed (Participants) | 214 | 220
titers
  rSBA-MenC at Month 3 | 1119.5 [926.4 to 1353.0] | 3200.5 [2737.7 to 3741.6]
  rSBA-MenC at Month 10: number analyzed (Participants) | 194 | 191
  rSBA-MenC at Month 10 | 131.1 [105.4 to 163.1] | 73.7 [56.9 to 95.3]
  rSBA-MenC at Month 11: number analyzed (Participants) | 199 | 196
  rSBA-MenC at Month 11 | 2653.8 [2225.5 to 3164.6] | 6028.4 [5183.4 to 7011.1]

7. Secondary Outcome: Number of Subjects With Anti-diphtheria (Anti-D) and Anti-tetanus (Anti-T) Antibodies Above the Cut-off.
Description: The anti-D and anti-T antibody cut-off was ≥ 0.1 international units per milliliter (IU/mL).
Time Frame: At Month 3, Month 10 and Month 11.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A Group | Infanrix Hexa Group
Number analyzed (Participants) | 216 | 223
Participants
  Anti-D at Month 3 | 215 | 222
  Anti-D at Month 10: number analyzed (Participants) | 197 | 195
  Anti-D at Month 10 | 143 | 169
  Anti-D at Month 11: number analyzed (Participants) | 200 | 196
  Anti-D at Month 11 | 200 | 196
  Anti-T at Month 3 | 216 | 223
  Anti-T at Month 10: number analyzed (Participants) | 197 | 195
  Anti-T at Month 10 | 189 | 176
  Anti-T at Month 11]: number analyzed (Participants) | 200 | 196
  Anti-T at Month 11] | 200 | 196

8. Secondary Outcome: Concentrations for Anti-T and Anti-D.
Description: Concentrations were expressed as geometric mean concentrations (GMCs). The reference cut-off value was ≥ 0.1 IU/mL.
Time Frame: At Month 3, Month 10 and Month 11.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | GSK2202083A Group | Infanrix Hexa Group
Number analyzed (Participants) | 216 | 223
IU/mL
  Anti-D at Month 3 | 0.936 [0.825 to 1.062] | 1.197 [1.069 to 1.340]
  Anti-D at Month 10: number analyzed (Participants) | 197 | 195
  Anti-D at Month 10 | 0.183 [0.159 to 0.211] | 0.241 [0.211 to 0.276]
  Anti-D at Month 11: number analyzed (Participants) | 200 | 196
  Anti-D at Month 11 | 4.538 [4.127 to 4.990] | 5.307 [4.862 to 5.793]
  Anti-T at Month 3 | 2.543 [2.332 to 2.774] | 1.380 [1.245 to 1.529]
  Anti-T at Month 10: number analyzed (Participants) | 197 | 195
  Anti-T at Month 10 | 0.458 [0.407 to 0.515] | 0.249 [0.219 to 0.282]
  Anti-T at Month 11: number analyzed (Participants) | 200 | 196
  Anti-T at Month 11 | 7.647 [7.063 to 8.279] | 4.720 [4.281 to 5.203]

9. Secondary Outcome: Number of Subjects With Anti-hepatitis B (Anti-HBs) Antibody Concentration Equal to or Above (≥) 10 and 100 Milli-International Units Per Milliliter (mIU/mL)
Description: A decrease in the specificity of the anti-HB enzyme-linked immunosorbent assay (ELISA) had been observed in some studies for low levels of antibody (10-100 mIU/mL). All the available blood samples initially tested with ELISA were re-tested using the Chemi Luminescence Immuno Assay (CLIA) approved by the US Food and Drug Administration (FDA). The table shows updated results following partial or complete retesting/reanalysis.
Time Frame: At Month 3, Month 10 and Month 11.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A Group | Infanrix Hexa Group
Number analyzed (Participants) | 207 | 216
Participants
  Anti-HBs ≥ 10 mIU/mL at Month 3 | 204 | 215
  Anti-HBs ≥ 10 mIU/mL at Month 10: number analyzed (Participants) | 197 | 195
  Anti-HBs ≥ 10 mIU/mL at Month 10 | 182 | 190
  Anti-HBs ≥ 10 mIU/mL at Month 11: number analyzed (Participants) | 196 | 196
  Anti-HBs ≥ 10 mIU/mL at Month 11 | 194 | 196
  Anti-HBs ≥ 100 mIU/mL at Month 3 | 190 | 207
  Anti-HBs ≥ 100 mIU/mL at Month 10: number analyzed (Participants) | 197 | 195
  Anti-HBs ≥ 100 mIU/mL at Month 10 | 118 | 146
  Anti-HBs ≥ 100 mIU/mL at Month 11: number analyzed (Participants) | 196 | 196
  Anti-HBs ≥ 100 mIU/mL at Month 11 | 187 | 194

10. Secondary Outcome: Concentrations for Anti-HBs.
Description: as for outcome 9
Time Frame: At Month 3, Month 10 and Month 11.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK2202083A Group | Infanrix Hexa Group
Number analyzed (Participants) | 207 | 216
mIU/mL
  Anti-HBs at Month 3 | 701.6 [578.4 to 851.1] | 897.8 [764.9 to 1053.9]
  Anti-HBs at Month 10: number analyzed (Participants) | 197 | 195
  Anti-HBs at Month 10 | 134.9 [107.6 to 169.2] | 212.8 [176.7 to 256.2]
  Anti-HBs at Month 11: number analyzed (Participants) | 196 | 196
  Anti-HBs at Month 11 | 3934.7 [3121.8 to 4959.3] | 4850.7 [4059.0 to 5796.9]

11. Secondary Outcome: Number of Subjects With Anti-poliovirus (Anti-polio) Types 1, 2 and 3 Above the Cut-off.
Description: The anti-polio 1, 2 and 3 antibody concentrations cut-off value was ≥ 1:8.
Time Frame: At Month 3, Month 10 and Month 11.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A Group | Infanrix Hexa Group
Number analyzed (Participants) | 196 | 208
Participants
  Anti-polio 1 at Month 3 | 168 | 183
  Anti-polio 1 at Month 10: number analyzed (Participants) | 183 | 188
  Anti-polio 1 at Month 10 | 82 | 98
  Anti-polio 1 at Month 11: number analyzed (Participants) | 191 | 189
  Anti-polio 1 at Month 11 | 182 | 186
  Anti-polio 2 at Month 3 | 159 | 160
  Anti-polio 2 at Month 10: number analyzed (Participants) | 183 | 188
  Anti-polio 2 at Month 10 | 87 | 96
  Anti-polio 2 at Month 11: number analyzed (Participants) | 191 | 189
  Anti-polio 2 at Month 11 | 188 | 186
  Anti-polio 3 at Month 3 | 169 | 188
  Anti-polio 3 at Month 10: number analyzed (Participants) | 183 | 188
  Anti-polio 3 at Month 10 | 96 | 108
  Anti-polio 3 at Month 11: number analyzed (Participants) | 191 | 189
  Anti-polio 3 at Month 11 | 188 | 185

12. Secondary Outcome: Titers for Anti-polio 1, 2 and 3.
Description: Titers were expressed as geometric mean titers (GMTs). The reference cut-off value was ≥ 1:8.
Time Frame: At Month 3, Month 10 and Month 11.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | GSK2202083A Group | Infanrix Hexa Group
Number analyzed (Participants) | 196 | 208
titers
  Anti-polio 1 at Month 3 | 37.5 [30.1 to 46.8] | 52.1 [42.1 to 64.5]
  Anti-polio 1 at Month 10: number analyzed (Participants) | 183 | 188
  Anti-polio 1 at Month 10 | 9.3 [7.8 to 10.9] | 11.2 [9.4 to 13.4]
  Anti-polio 1 at Month 11: number analyzed (Participants) | 191 | 189
  Anti-polio 1 at Month 11 | 268.4 [216.5 to 332.7] | 313.7 [258.7 to 380.4]
  Anti-polio 2 at Month 3 | 28.1 [22.6 to 35.0] | 30.6 [24.5 to 38.2]
  Anti-polio 2 at Month 10: number analyzed (Participants) | 183 | 188
  Anti-polio 2 at Month 10 | 10.0 [8.4 to 11.9] | 10.5 [8.8 to 12.4]
  Anti-polio 2 at Month 11: number analyzed (Participants) | 191 | 189
  Anti-polio 2 at Month 11 | 379.0 [311.0 to 461.9] | 429.2 [357.6 to 515.2]
  Anti-polio 3 at Month 3 | 70.0 [54.0 to 90.7] | 91.9 [71.8 to 117.6]
  Anti-polio 3 at Month 10: number analyzed (Participants) | 183 | 188
  Anti-polio 3 at Month 10 | 13.0 [10.7 to 15.9] | 15.1 [12.4 to 18.4]
  Anti-polio 3 at Month 11: number analyzed (Participants) | 191 | 189
  Anti-polio 3 at Month 11 | 506.5 [407.9 to 628.9] | 541.9 [443.6 to 661.9]

13. Secondary Outcome: Number Subjects With Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Haemagglutinin (Anti-FHA) and Anti-pertactin (Anti-PRN) Above the Cut-off.
Description: The reference cut-off for anti-PT, anti-FHA and anti-PRN antibody concentrations was ≥ 5 enzyme-linked immunosorbent assay (ELISA) units per milliliters (EL.U/mL).
Time Frame: At Month 3, Month 10 and Month 11.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A Group | Infanrix Hexa Group
Number analyzed (Participants) | 217 | 223
Participants
  Anti-PT at Month 3 | 217 | 223
  Anti-PT at Month 10: number analyzed (Participants) | 193 | 194
  Anti-PT at Month 10 | 136 | 153
  Anti-PT at Month 11: number analyzed (Participants) | 200 | 196
  Anti-PT at Month 11 | 199 | 195
  Anti-FHA at Month 3: number analyzed (Participants) | 216 | 222
  Anti-FHA at Month 3 | 216 | 222
  Anti-FHA at Month 10: number analyzed (Participants) | 197 | 196
  Anti-FHA at Month 10 | 196 | 195
  Anti-FHA at Month 11: number analyzed (Participants) | 199 | 196
  Anti-FHA at Month 11 | 199 | 196
  Anti-PRN at Month 3 | 216 | 222
  Anti-PRN at Month 10: number analyzed (Participants) | 197 | 196
  Anti-PRN at Month 10 | 129 | 142
  Anti-PRN at Month 11: number analyzed (Participants) | 200 | 198
  Anti-PRN at Month 11 | 200 | 198

14. Secondary Outcome: Concentrations for Anti-PT, Anti-FHA and Anti-PRN.
Description: Concentrations were expressed as geometric mean concentrations (GMCs). The reference cut-off value was ≥ 5 EL.U/mL.
Time Frame: At Month 3, Month 10 and Month 11.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | GSK2202083A Group | Infanrix Hexa Group
Number analyzed (Participants) | 217 | 223
EL.U/mL
  Anti-PT at Month 3 | 47.4 [43.3 to 51.9] | 49.3 [45.6 to 53.3]
  Anti-PT at Month 10: number analyzed (Participants) | 193 | 194
  Anti-PT at Month 10 | 8.0 [7.0 to 9.1] | 8.3 [7.4 to 9.3]
  Anti-PT at Month 11: number analyzed (Participants) | 200 | 196
  Anti-PT at Month 11 | 74.9 [67.2 to 83.5] | 86.1 [77.8 to 95.4]
  Anti-FHA at Month 3: number analyzed (Participants) | 216 | 222
  Anti-FHA at Month 3 | 165.8 [151.5 to 181.5] | 172.3 [157.9 to 188.1]
  Anti-FHA at Month 10: number analyzed (Participants) | 197 | 196
  Anti-FHA at Month 10 | 37.8 [33.3 to 43.0] | 39.7 [35.3 to 44.6]
  Anti-FHA at Month 11: number analyzed (Participants) | 199 | 196
  Anti-FHA at Month 11 | 429.6 [388.4 to 475.0] | 451.2 [413.7 to 492.1]
  Anti-PRN at Month 3 | 66.2 [56.9 to 77.0] | 74.5 [64.7 to 85.7]
  Anti-PRN at Month 10: number analyzed (Participants) | 197 | 196
  Anti-PRN at Month 10 | 9.1 [7.7 to 10.8] | 11.0 [9.3 to 13.1]
  Anti-PRN at Month 11: number analyzed (Participants) | 200 | 198
  Anti-PRN at Month 11 | 218.0 [188.5 to 252.2] | 242.9 [216.1 to 273.1]

15. Secondary Outcome: Number of Subjects With a Booster Response to Anti-PT, Anti-FHA and Anti-PRN.
Description: Booster response defined as: for initially seronegative subjects, antibody concentration ≥ 5 EL.U/mL at Month 11; for initially seropositive subjects: antibody concentration at Month 11 ≥ 2 fold the pre-vaccination antibody concentration
Time Frame: At Month 11.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A Group | Infanrix Hexa Group
Number analyzed (Participants) | 193 | 193
Participants
  Anti-FHA: number analyzed (Participants) | 191 | 190
  Anti-FHA | 183 | 185
  Anti-PRN | 191 | 190
  Anti-PT: number analyzed (Participants) | 189 | 189
  Anti-PT | 185 | 186

16. Secondary Outcome: Number of Subjects With Anti-pneumococcal (Anti-PNE) Serotypes Above the Cut-offs.
Description: The anti-PNE antibody concentrations reference cut-offs were ≥ 0.2 and ≥ 0.05 micrograms per milliliter (µg/mL). The anti-PNE serotypes assessed were 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F.
Time Frame: At Month 3 and Month 11
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A Group | Infanrix Hexa Group
Number analyzed (Participants) | 87 | 94
Participants
  Anti-PNE 1 at Month 3 ≥ 0.2 | 86 | 94
  Anti-PNE 1 at Month 11 ≥ 0.2: number analyzed (Participants) | 86 | 83
  Anti-PNE 1 at Month 11 ≥ 0.2 | 86 | 83
  Anti-PNE 3 at Month 3 ≥ 0.2: number analyzed (Participants) | 83 | 93
  Anti-PNE 3 at Month 3 ≥ 0.2 | 82 | 93
  Anti-PNE 3 at Month 11 ≥ 0.2: number analyzed (Participants) | 86 | 83
  Anti-PNE 3 at Month 11 ≥ 0.2 | 83 | 83
  Anti-PNE 4 at Month 3 ≥ 0.2: number analyzed (Participants) | 82 | 94
  Anti-PNE 4 at Month 3 ≥ 0.2 | 78 | 93
  Anti-PNE 4 at Month 11 ≥ 0.2: number analyzed (Participants) | 86 | 83
  Anti-PNE 4 at Month 11 ≥ 0.2 | 85 | 83
  Anti-PNE 5 at Month 3 ≥ 0.2: number analyzed (Participants) | 80 | 91
  Anti-PNE 5 at Month 3 ≥ 0.2 | 75 | 89
  Anti-PNE 5 at Month 11 ≥ 0.2: number analyzed (Participants) | 86 | 83
  Anti-PNE 5 at Month 11 ≥ 0.2 | 86 | 83
  Anti-PNE 6A at Month 3 ≥ 0.2: number analyzed (Participants) | 80 | 92
  Anti-PNE 6A at Month 3 ≥ 0.2 | 70 | 86
  Anti-PNE 6A at Month 11 ≥ 0.2: number analyzed (Participants) | 86 | 83
  Anti-PNE 6A at Month 11 ≥ 0.2 | 84 | 83
  Anti-PNE 6B at Month 3 ≥ 0.2: number analyzed (Participants) | 80 | 92
  Anti-PNE 6B at Month 3 ≥ 0.2 | 20 | 27
  Anti-PNE 6B at Month 11 ≥ 0.2: number analyzed (Participants) | 86 | 83
  Anti-PNE 6B at Month 11 ≥ 0.2 | 83 | 82
  Anti-PNE 7F at Month 3 ≥ 0.2: number analyzed (Participants) | 84 | 93
  Anti-PNE 7F at Month 3 ≥ 0.2 | 83 | 93
  Anti-PNE 7F at Month 11 ≥ 0.2: number analyzed (Participants) | 86 | 83
  Anti-PNE 7F at Month 11 ≥ 0.2 | 86 | 83
  Anti-PNE 9V at Month 3 ≥ 0.2: number analyzed (Participants) | 82 | 91
  Anti-PNE 9V at Month 3 ≥ 0.2 | 77 | 89
  Anti-PNE 9V at Month 11 ≥ 0.2: number analyzed (Participants) | 86 | 83
  Anti-PNE 9V at Month 11 ≥ 0.2 | 85 | 83
  Anti-PNE 14 at Month 3 ≥ 0.2: number analyzed (Participants) | 85 | 93
  Anti-PNE 14 at Month 3 ≥ 0.2 | 85 | 92
  Anti-PNE 14 at Month 11 ≥ 0.2: number analyzed (Participants) | 86 | 83
  Anti-PNE 14 at Month 11 ≥ 0.2 | 86 | 82
  Anti-PNE 18C at Month 3 ≥ 0.2: number analyzed (Participants) | 83 | 93
  Anti-PNE 18C at Month 3 ≥ 0.2 | 79 | 89
  Anti-PNE 18C at Month 11 ≥ 0.2: number analyzed (Participants) | 86 | 83
  Anti-PNE 18C at Month 11 ≥ 0.2 | 86 | 83
  Anti-PNE 19A at Month 3 ≥ 0.2: number analyzed (Participants) | 83 | 93
  Anti-PNE 19A at Month 3 ≥ 0.2 | 74 | 91
  Anti-PNE 19A at Month 11 ≥ 0.2: number analyzed (Participants) | 86 | 83
  Anti-PNE 19A at Month 11 ≥ 0.2 | 85 | 83
  Anti-PNE 19F at Month 3 ≥ 0.2: number analyzed (Participants) | 81 | 92
  Anti-PNE 19F at Month 3 ≥ 0.2 | 79 | 92
  Anti-PNE 19F at Month 11 ≥ 0.2: number analyzed (Participants) | 85 | 82
  Anti-PNE 19F at Month 11 ≥ 0.2 | 84 | 82
  Anti-PNE 23F at Month 3 ≥ 0.2: number analyzed (Participants) | 77 | 92
  Anti-PNE 23F at Month 3 ≥ 0.2 | 52 | 76
  Anti-PNE 23F at Month 11 ≥ 0.2: number analyzed (Participants) | 86 | 83
  Anti-PNE 23F at Month 11 ≥ 0.2 | 84 | 82
  Anti-PNE 1 at Month 3 ≥ 0.05 | 87 | 94
  Anti-PNE 1 at Month 11 ≥ 0.05: number analyzed (Participants) | 86 | 83
  Anti-PNE 1 at Month 11 ≥ 0.05 | 86 | 83
  Anti-PNE 3 at Month 3 ≥ 0.05: number analyzed (Participants) | 83 | 93
  Anti-PNE 3 at Month 3 ≥ 0.05 | 83 | 93
  Anti-PNE 3 at Month 11 ≥ 0.05: number analyzed (Participants) | 86 | 83
  Anti-PNE 3 at Month 11 ≥ 0.05 | 85 | 83
  Anti-PNE 4 at Month 3 ≥ 0.05: number analyzed (Participants) | 82 | 94
  Anti-PNE 4 at Month 3 ≥ 0.05 | 82 | 94
  Anti-PNE 4 at Month 11 ≥ 0.05: number analyzed (Participants) | 86 | 83
  Anti-PNE 4 at Month 11 ≥ 0.05 | 86 | 83
  Anti-PNE 5 at Month 3 ≥ 0.05: number analyzed (Participants) | 80 | 91
  Anti-PNE 5 at Month 3 ≥ 0.05 | 79 | 91
  Anti-PNE 5 at Month 11 ≥ 0.05: number analyzed (Participants) | 86 | 83
  Anti-PNE 5 at Month 11 ≥ 0.05 | 86 | 83
  Anti-PNE 6A at Month 3 ≥ 0.05: number analyzed (Participants) | 80 | 92
  Anti-PNE 6A at Month 3 ≥ 0.05 | 79 | 91
  Anti-PNE 6A at Month 11 ≥ 0.05: number analyzed (Participants) | 86 | 83
  Anti-PNE 6A at Month 11 ≥ 0.05 | 86 | 83
  Anti-PNE 6B at Month 3 ≥ 0.05: number analyzed (Participants) | 80 | 92
  Anti-PNE 6B at Month 3 ≥ 0.05 | 54 | 72
  Anti-PNE 6B at Month 11 ≥ 0.05: number analyzed (Participants) | 86 | 83
  Anti-PNE 6B at Month 11 ≥ 0.05 | 85 | 83
  Anti-PNE 7F at Month 3 ≥ 0.05: number analyzed (Participants) | 84 | 93
  Anti-PNE 7F at Month 3 ≥ 0.05 | 84 | 93
  Anti-PNE 7F at Month 11 ≥ 0.05: number analyzed (Participants) | 86 | 83
  Anti-PNE 7F at Month 11 ≥ 0.05 | 86 | 83
  Anti-PNE 9V at Month 3 ≥ 0.05: number analyzed (Participants) | 82 | 91
  Anti-PNE 9V at Month 3 ≥ 0.05 | 80 | 91
  Anti-PNE 9V at Month 11 ≥ 0.05: number analyzed (Participants) | 86 | 83
  Anti-PNE 9V at Month 11 ≥ 0.05 | 86 | 83
  Anti-PNE 14 at Month 3 ≥ 0.05: number analyzed (Participants) | 85 | 93
  Anti-PNE 14 at Month 3 ≥ 0.05 | 85 | 93
  Anti-PNE 14 at Month 11 ≥ 0.05: number analyzed (Participants) | 86 | 83
  Anti-PNE 14 at Month 11 ≥ 0.05 | 86 | 83
  Anti-PNE 18C at Month 3 ≥ 0.05: number analyzed (Participants) | 83 | 93
  Anti-PNE 18C at Month 3 ≥ 0.05 | 83 | 93
  Anti-PNE 18C at Month 11 ≥ 0.05: number analyzed (Participants) | 86 | 83
  Anti-PNE 18C at Month 11 ≥ 0.05 | 86 | 83
  Anti-PNE 19A at Month 3 ≥ 0.05: number analyzed (Participants) | 83 | 93
  Anti-PNE 19A at Month 3 ≥ 0.05 | 83 | 93
  Anti-PNE 19A at Month 11 ≥ 0.05: number analyzed (Participants) | 86 | 83
  Anti-PNE 19A at Month 11 ≥ 0.05 | 86 | 83
  Anti-PNE 19F at Month 3 ≥ 0.05: number analyzed (Participants) | 81 | 92
  Anti-PNE 19F at Month 3 ≥ 0.05 | 81 | 92
  Anti-PNE 19F at Month 11 ≥ 0.05: number analyzed (Participants) | 85 | 82
  Anti-PNE 19F at Month 11 ≥ 0.05 | 85 | 82
  Anti-PNE 23F at Month 3 ≥ 0.05: number analyzed (Participants) | 77 | 92
  Anti-PNE 23F at Month 3 ≥ 0.05 | 73 | 89
  Anti-PNE 23F at Month 11 ≥ 0.05: number analyzed (Participants) | 86 | 83
  Anti-PNE 23F at Month 11 ≥ 0.05 | 85 | 82

17. Secondary Outcome: Concentrations for Anti-PNE Serotypes.
Description: Concentrations were expressed as geometric mean concentreations (GMCs). The reference cut-off value was ≥ 0.2 µg/mL.
Time Frame: At Month 3 and Month 11
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | GSK2202083A Group | Infanrix Hexa Group
Number analyzed (Participants) | 87 | 94
µg/mL
  Anti-PNE 1 at Month 3 ≥ 0.2 | 1.66 [1.37 to 2.00] | 1.89 [1.59 to 2.25]
  Anti-PNE 1 at Month 11 ≥ 0.2: number analyzed (Participants) | 86 | 83
  Anti-PNE 1 at Month 11 ≥ 0.2 | 4.99 [4.13 to 6.02] | 4.79 [4.12 to 5.56]
  Anti-PNE 3 at Month 3 ≥ 0.2: number analyzed (Participants) | 83 | 93
  Anti-PNE 3 at Month 3 ≥ 0.2 | 1.16 [0.99 to 1.35] | 1.15 [1.02 to 1.30]
  Anti-PNE 3 at Month 11 ≥ 0.2: number analyzed (Participants) | 86 | 83
  Anti-PNE 3 at Month 11 ≥ 0.2 | 1.74 [1.41 to 2.16] | 1.82 [1.54 to 2.15]
  Anti-PNE 4 at Month 3 ≥ 0.2: number analyzed (Participants) | 82 | 94
  Anti-PNE 4 at Month 3 ≥ 0.2 | 1.40 [1.14 to 1.73] | 1.55 [1.32 to 1.82]
  Anti-PNE 4 at Month 11 ≥ 0.2: number analyzed (Participants) | 86 | 83
  Anti-PNE 4 at Month 11 ≥ 0.2 | 4.19 [3.46 to 5.06] | 4.43 [3.77 to 5.21]
  Anti-PNE 5 at Month 3 ≥ 0.2: number analyzed (Participants) | 80 | 91
  Anti-PNE 5 at Month 3 ≥ 0.2 | 1.83 [1.38 to 2.43] | 2.17 [1.76 to 2.68]
  Anti-PNE 5 at Month 11 ≥ 0.2: number analyzed (Participants) | 86 | 83
  Anti-PNE 5 at Month 11 ≥ 0.2 | 6.68 [5.47 to 8.17] | 6.75 [5.67 to 8.02]
  Anti-PNE 6A at Month 3 ≥ 0.2: number analyzed (Participants) | 80 | 92
  Anti-PNE 6A at Month 3 ≥ 0.2 | 1.06 [0.82 to 1.39] | 1.20 [0.98 to 1.48]
  Anti-PNE 6A at Month 11 ≥ 0.2: number analyzed (Participants) | 86 | 83
  Anti-PNE 6A at Month 11 ≥ 0.2 | 7.34 [5.87 to 9.16] | 7.96 [6.95 to 9.11]
  Anti-PNE 6B at Month 3 ≥ 0.2: number analyzed (Participants) | 80 | 92
  Anti-PNE 6B at Month 3 ≥ 0.2 | 0.09 [0.07 to 0.12] | 0.12 [0.09 to 0.15]
  Anti-PNE 6B at Month 11 ≥ 0.2: number analyzed (Participants) | 86 | 83
  Anti-PNE 6B at Month 11 ≥ 0.2 | 2.23 [1.68 to 2.97] | 2.78 [2.23 to 3.46]
  Anti-PNE 7F at Month 3 ≥ 0.2: number analyzed (Participants) | 84 | 93
  Anti-PNE 7F at Month 3 ≥ 0.2 | 2.72 [2.30 to 3.21] | 2.75 [2.44 to 3.10]
  Anti-PNE 7F at Month 11 ≥ 0.2: number analyzed (Participants) | 86 | 83
  Anti-PNE 7F at Month 11 ≥ 0.2 | 6.67 [5.82 to 7.65] | 6.47 [5.68 to 7.38]
  Anti-PNE 9V at Month 3 ≥ 0.2: number analyzed (Participants) | 82 | 91
  Anti-PNE 9V at Month 3 ≥ 0.2 | 1.36 [1.02 to 1.82] | 1.42 [1.17 to 1.74]
  Anti-PNE 9V at Month 11 ≥ 0.2: number analyzed (Participants) | 86 | 83
  Anti-PNE 9V at Month 11 ≥ 0.2 | 6.12 [4.99 to 7.50] | 6.80 [5.78 to 8.00]
  Anti-PNE 14 at Month 3 ≥ 0.2: number analyzed (Participants) | 85 | 93
  Anti-PNE 14 at Month 3 ≥ 0.2 | 3.03 [2.42 to 3.80] | 2.96 [2.33 to 3.76]
  Anti-PNE 14 at Month 11 ≥ 0.2: number analyzed (Participants) | 86 | 83
  Anti-PNE 14 at Month 11 ≥ 0.2 | 10.41 [8.56 to 12.65] | 7.50 [6.03 to 9.34]
  Anti-PNE 18C at Month 3 ≥ 0.2: number analyzed (Participants) | 83 | 93
  Anti-PNE 18C at Month 3 ≥ 0.2 | 1.81 [1.40 to 2.34] | 2.08 [1.72 to 2.51]
  Anti-PNE 18C at Month 11 ≥ 0.2: number analyzed (Participants) | 86 | 83
  Anti-PNE 18C at Month 11 ≥ 0.2 | 6.20 [5.06 to 7.59] | 5.91 [4.97 to 7.02]
  Anti-PNE 19A at Month 3 ≥ 0.2: number analyzed (Participants) | 83 | 93
  Anti-PNE 19A at Month 3 ≥ 0.2 | 1.05 [0.81 to 1.36] | 1.30 [1.10 to 1.54]
  Anti-PNE 19A at Month 11 ≥ 0.2: number analyzed (Participants) | 86 | 83
  Anti-PNE 19A at Month 11 ≥ 0.2 | 5.73 [4.55 to 7.20] | 5.22 [4.26 to 6.41]
  Anti-PNE 19F at Month 3 ≥ 0.2: number analyzed (Participants) | 81 | 92
  Anti-PNE 19F at Month 3 ≥ 0.2 | 2.82 [2.25 to 3.53] | 3.36 [2.83 to 3.98]
  Anti-PNE 19F at Month 11 ≥ 0.2: number analyzed (Participants) | 85 | 82
  Anti-PNE 19F at Month 11 ≥ 0.2 | 5.47 [4.36 to 6.86] | 5.70 [4.81 to 6.75]
  Anti-PNE 23F at Month 3 ≥ 0.2: number analyzed (Participants) | 77 | 92
  Anti-PNE 23F at Month 3 ≥ 0.2 | 0.40 [0.29 to 0.54] | 0.54 [0.43 to 0.68]
  Anti-PNE 23F at Month 11 ≥ 0.2: number analyzed (Participants) | 86 | 83
  Anti-PNE 23F at Month 11 ≥ 0.2 | 4.38 [3.33 to 5.77] | 4.51 [3.57 to 5.69]

18. Secondary Outcome: Number of Subjects With Anti-PRP and rSBA-MenC Fold Increase Distribution.
Description: The fold increase distribution cut-offs were: ≥2, ≥4, ≥6, ≥8 and ≥10.
Time Frame: At Month 11.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A Group | Infanrix Hexa Group
Number analyzed (Participants) | 197 | 193
Participants
  Anti-PRP ≥2 | 195 | 189
  Anti-PRP ≥4 | 191 | 186
  Anti-PRP ≥6 | 189 | 176
  Anti-PRP ≥8 | 179 | 170
  Anti-PRP ≥10 | 173 | 166
  rSBA-MenC ≥2: number analyzed (Participants) | 193 | 189
  rSBA-MenC ≥2 | 189 | 185
  rSBA-MenC ≥4: number analyzed (Participants) | 193 | 189
  rSBA-MenC ≥4 | 177 | 185
  rSBA-MenC ≥6: number analyzed (Participants) | 193 | 189
  rSBA-MenC ≥6 | 160 | 182
  rSBA-MenC ≥8: number analyzed (Participants) | 193 | 189
  rSBA-MenC ≥8 | 148 | 180
  rSBA-MenC ≥10: number analyzed (Participants) | 193 | 189
  rSBA-MenC ≥10 | 135 | 178

19. Secondary Outcome: Number of Subjects Reporting Any Solicited Local Symptoms.
Description: Solicited local symptoms assessed were pain, redness and swelling. Any = occurrence of any local symptom regardless of intensity grade.
Time Frame: During the 8-day (Days 0-7) post-vaccination period
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one vaccine administration documented and the symptom sheet completed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A Group | Infanrix Hexa Group
Number analyzed (Participants) | 238 | 241
Participants
  Any pain | 155 | 181
  Any redness | 171 | 183
  Any swelling | 147 | 163

20. Secondary Outcome: Number of Subjects Reporting Any Solicited General Symptoms.
Description: Solicited local symptoms assessed were drowsiness, irritability/fussiness, loss of appetite and fever [axillary temperature above (≥) 37.5 degrees Celsius (°C)]. Any = occurrence of any local symptom regardless of intensity grade.
Time Frame: During the 8-day (Days 0-7) post-vaccination period
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A Group | Infanrix Hexa Group
Number analyzed (Participants) | 238 | 241
Participants
  Any drowsiness | 188 | 190
  Any irritability | 208 | 207
  Any loss of appetite | 169 | 154
  Any fever | 165 | 167

21. Secondary Outcome: Number of Subjects Reporting Any Unsolicited Adverse Events (AEs).
Description: An unsolicited AE is any AE (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any = occurrence of an AE regardless of intensity grade or relationship to study vaccination.
Time Frame: Within the 31-day (Days 0-30) follow up period after vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one vaccine administration documented.
Measure: Number; unit: Subjects
Arm/Group | GSK2202083A Group | Infanrix Hexa Group
Number analyzed (Participants) | 238 | 242
Subjects | 148 | 158

22. Secondary Outcome: Number of Subjects Reporting Any Serious Adverse Events (SAEs).
Description: SAEs assessed include medical occurrences that results in death, are life threatening, require hospitalization or prolongation of hospitalization, results in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subjects. Any SAE = any SAE regardless of assessment of relationship to study vaccination.
Time Frame: During the entire study period (Month 0 to Month 11)
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A Group | Infanrix Hexa Group
Number analyzed (Participants) | 238 | 242
Participants | 12 | 15

ADVERSE EVENTS:
Time Frame: Solicited symptoms: 8-day (Days 0-7) follow-up period after vaccination; unsolicited AEs: 31-day (Days 0-30) follow-up period after vaccination; SAEs: during the entire study period (Months 0-11).
Description: For solicited local and general symptoms, the number of participants at risk included those from Total Vaccinated cohort who had the symptom sheet completed.
Arm/Group | GSK2202083A Group | Infanrix Hexa Group
All-Cause Mortality (participants affected / at risk) | 0/238 | 0/242
Serious Adverse Events (participants affected / at risk) | 12/238 | 15/242
Other Adverse Events (participants affected / at risk) | 232/238 | 237/242
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2202083A Group (N=238) | Infanrix Hexa Group (N=242)
Concussion (Injury, poisoning and procedural complications) | 0 | 3
Gastroenteritis (Infections and infestations) | 1 | 1
Accidental drug intake by child (Injury, poisoning and procedural complications) | 1 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cow's milk intolerance (Metabolism and nutrition disorders) | 1 | 0
Croup infectious (Infections and infestations) | 0 | 1
Crying (General disorders) | 1 | 0
Gastroenteritis adenovirus (Infections and infestations) | 0 | 1
Gastroenteritis norovirus (Infections and infestations) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Otitis media (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Rash (Infections and infestations) | 0 | 1
Sandifer's syndrome (Gastrointestinal disorders) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | GSK2202083A Group (N=238) | Infanrix Hexa Group (N=242)
Rhinitis (Infections and infestations) | 31 | 27
Upper respiratory tract infection (Infections and infestations) | 20 | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 19 | 14
Diarrhoea (Gastrointestinal disorders) | 12 | 17
Nasopharyngitis (Infections and infestations) | 10 | 16
Vomiting (Gastrointestinal disorders) | 9 | 14
Pain (General disorders) | 155 | 181/241 — This solicited local symptom was only collected from subjects with their symptom sheets completed.
Redness (General disorders) | 171 | 183/241 — This solicited local symptom was only collected from subjects with their symptom sheets completed.
Swelling (General disorders) | 147 | 163/241 — This solicited local symptom was only collected from subjects with their symptom sheets completed.
Drowsiness (General disorders) | 188 | 190/241 — This solicited general symptom was only collected from subjects with their symptom sheets completed.
Irritability (General disorders) | 208 | 207/241 — This solicited general symptom was only collected from subjects with their symptom sheets completed.
Loss of appetite (General disorders) | 169 | 154/241 — This solicited general symptom was only collected from subjects with their symptom sheets completed.
Temperature (General disorders) | 165 | 167/241 — This solicited general symptom was only collected from subjects with their symptom sheets completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.